CLINICAL TRIAL: NCT03949374
Title: A 8-week, Single Center, Randomized, Open-label, Parallel-group, Non-inferiority Clinical Trial to Evaluate Efficacy and Safety of ROVASRO 10mg Versus CRESTOR 10mg in Hypercholesterolemic Patients
Brief Title: Clinical Trial to Evaluate Efficacy and Safety of ROVASRO 10mg Versus CRESTOR 10mg in Hypercholesterolemic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0730
Record Dates: First submitted 2019-05-03; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Hypercholesterolemia; Dyslipidemias
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: 10mg of the generic formulation (rosuvastatin, ROVASRO®) versus 10mg of the reference formulation (rosuvastatin, CRESTOR®)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10mg of the generic formulation (rosuvastatin, ROVASRO®) (Active Comparator): Taking 10mg of the generic formulation (rosuvastatin, ROVASRO®)
  Interventions: Drug: ROVASRO, generic formulation of rosuvastatin
- 10mg of the reference formulation (rosuvastatin, CRESTOR®) (Active Comparator): Taking 10mg of the reference formulation (rosuvastatin, CRESTOR®)
  Interventions: Drug: CRESTOR, reference formulation of rosuvastatin

INTERVENTIONS:
Drug: CRESTOR, reference formulation of rosuvastatin — Use of ROVASRO for hypercholesterolemia
  Arms: 10mg of the reference formulation (rosuvastatin, CRESTOR®)
Drug: ROVASRO, generic formulation of rosuvastatin — Use of CRESTOR for hypercholesterolemia
  Arms: 10mg of the generic formulation (rosuvastatin, ROVASRO®)

SUMMARY:
This 8 weeks, prospective, single center, randomized, open-label, parallel-group, non-inferiority study was performed from October 2015 to April 2018. This study as designed to evaluate the efficacy and safety of 10mg of the generic formulation (rosuvastatin, ROVASRO®) compared to the reference formulation (rosuvastatin, CRESTOR®) in patients with primary hypercholesterolemia and complex dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged between 19 and 80 years old.
2. The following patients who belong to the low-risk group to the very-high risk group according to 2015 Korean guidelines for the management of dyslipidemia (Committee, KCJ 2016).

   * Very high risk group (coronary artery disease, ischemic stroke, peripheral vascular disease) were not receiving lipid-lowering agents (statins) within 4 weeks of the screening, regardless of LDL-C levels
   * High risk group (carotid artery disease, abnormal aneurysm, diabetes)* : LDL-C ≥ 100 mg/dl
   * Moderate risk group (2 or more major risk factors)* : LDL-C ≥ 130 mg/dl
   * Low risk group (less than 1 major risk factors)* : LDL-C ≥ 160 mg/dl

     * If the patients taka a lipid-lowering agents (statin) within 4 weeks of screening, enrolled them after wash-out for 4 weeks or more.
3. Patients who voluntarily participated in the trial and obtained document consent.

Exclusion Criteria:

1. a history of acute arterial disease (patients with unstable angina myocardial infarction, transient ischemic attack, cerebrovascular disease, coronary artery bypass graft or percutaneous transluminal coronary angioplasty within 3 months prior to study enrollment)
2. uncontrolled hypertension (systolic blood pressure ≥180mmHg or diastolic blood pressure ≥100mmHg)
3. uncontrolled diabetes (hemoglobin A1c ≥9% or fasting glucose ≥160mg/dl)
4. uncontrolled thyroid dysfunction (thyroid stimulation hormone ≥1.5 times the upper limits of normal (ULN))
5. usage of antihyperlipidemic drugs (bile acid sequestrants, fibrates, niacin, etc.) within 4 weeks before enrollment
6. a history of myopathy, rhabdomyolysis or elevated serum creatinine kinase (CK) more than 2 times the ULN
7. chronic kidney disease (serum creatinine ≥2 times the ULN)
8. elevated liver enzymes (aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2 times the ULN)
9. a history of drug or alcohol abuse
10. a history of gastrointestinal surgery or gastrointestinal tract disorders
11. hypersensitivity to the components of this drug
12. those who disagree with contraception
13. pregnancy and/or lactation.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage change in the level of LDL-C | 8 weeks after treatment
  Percentage change in the level of low-density lipoprotein-cholesterol (LDL-C)(mg/dL) from baseline to week 8 of drug treatment.
Target achievement rate in the level of LDL-C | 8 weeks after treatment
  Target achievement rate in the level of LDL-C from baseline to week 8 of drug treatment The LDL-C targets were defined as <70 mg/dL for the very high risk group, <100 mg/dL for the high risk group, <130 mg/dL for the moderate risk group, and <160 mg/dL for the low risk group (Committee. KCJ 2016).

SECONDARY OUTCOMES:
Change in biochemical parameters : total cholesterol (mg/dL) | 8 weeks after treatment
  Percentage changes in total cholesterol (mg/dL).
Change in biochemical parameters : triglyceride (mg/dL) | 8 weeks after treatment
  Percentage changes in triglyceride (mg/dL).
Change in biochemical parameters : high-density lipoprotein-cholesterol(HDL-C)(mg/dL) | 8 weeks after treatment
  Percentage changes in high-density lipoprotein-cholesterol(HDL-C)(mg/dL).
Change in biochemical parameters : apolipoprotein B(mg/dL) | 8 weeks after treatment
  Percentage changes in apolipoprotein B(mg/dL).
Change in biochemical parameters : apolipoprotein A1(mg/dL) | 8 weeks after treatment
  Percentage changes in apolipoprotein A1(mg/dL).
Change in biochemical parameters : high sensitivity C-reactive protein (hsCRP)(mg/L) | 8 weeks after treatment
  Percentage changes in high sensitivity C-reactive protein (hsCRP)(mg/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Cardiovascular Center, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim H, Lee CJ, Choi D, Kim BK, Kim IC, Kim JS, Ahn CM, Hong GR, Cho IJ, Shim CY, Lee SH. Lipid-Lowering Efficacy and Safety of a New Generic Rosuvastatin in Koreans: an 8-Week Randomized Comparative Study with a Proprietary Rosuvastatin. J Lipid Atheroscler. 2020 May;9(2):283-290. doi: 10.12997/jla.2020.9.2.283. Epub 2020 Mar 6. PMID 32821737